CLINICAL TRIAL: NCT02380937
Title: Radio Frequency Ablation for Atrial Flutter With Magnetic Resonance Guidance and Tracking: Pilot Study Using a Combination Imricor and Philips Interventional System
Brief Title: Radio Frequency Ablation for Atrial Flutter With Magnetic Resonance Guidance and Tracking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely on 05May 2015 because of the unavailability of study devices.
Sponsor: University of Leipzig (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other); Philips Healthcare (Industry); Imricor Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104/14-ff
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2015-11

CONDITIONS: Atrial Flutter
Keywords: real-time MRI; electrophysiology study; atrial flutter; ablation; active tracking
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ablation for typical atrial flutter (Experimental): This group receives an MR-guide ablation for atrial flutter with the study device (catheter)
  Interventions: Procedure: ablation for typical atrial flutter; Device: Vision Ablation Catheter

INTERVENTIONS:
Procedure: ablation for typical atrial flutter — ablation for typical atrial flutter
Device: Vision Ablation Catheter

SUMMARY:
The Radio Frequency Ablation for Atrial Flutter with Magnetic Resonance Guidance and Tracking Pilot Study (hereafter referred to as "pilot study") is a prospective, non- randomized, single-center, pilot study. The purpose of this clinical study is to evaluate the safety and performance of the Imricor Medical Systems, Inc. (Imricor) Vision Ablation Catheter when used with related accessories for the treatment of type I atrial flutter. The Vision Ablation Catheter and its accessories have been designed for use under fluoroscopic or magnetic resonance guidance.

DETAILED DESCRIPTION:
An objective of the study is to perform the entire ablation procedure from subject preparation through confirmation of bidirectional conduction block entirely under magnetic resonance guidance. However, at the investigator's discretion, the preparation of the subject may occur in a conventional electrophysiology laboratory followed by transferring the patient to the magnetic resonance suite for the ablation procedure. Additionally, if bidirectional conduction block is not achieved within 90 minutes from the initial catheter placement, the subject may be transferred from the magnetic resonance suite to a conventional electrophysiology lab to complete the procedure. Clinical success is bidirectional conduction block regardless of the environment within which the ablation occurs.

The study will be conducted at a single center, Herzzentrum Leipzig University Hospital, in Germany, and a maximum of 30 subjects meeting inclusion/exclusion criteria will participate in the study. This study requires the use of investigational products from two independent manufacturers: Imricor and Philips. Imricor has developed the ablation catheter with related accessories, introducers, and recording system. Philips has developed an image guidance and mapping system that is compatible with the Imricor products. The Vision Ablation Catheter will be used in conjunction with the following investigational products: Vision Ablation Catheter Cable Set (accessory sterile cable), Vision Hemostasis Introducer, Vision Dual-Deflect Sheath, Horizon recording system, and the interventional MRI Suite (iSuite) image guidance and mapping system. With the exception of iSuite, which is manufactured by Philips, Imricor will provide all investigational devices used in the study. Each procedure will utilize the following two single-use products: two Vision Ablation Catheters and an accessory Catheter Cable set. At the discretion of the investigator, Vision Hemostasis Introducers may be used for femoral access and a Vision Dual- Deflect Sheath and may be used in conjunction with the Vision Ablation Catheter Cable Set. Ablation for the treatment of arrhythmia is an inherently complex procedure. Use of the investigational products listed above under magnetic resonance guidance is a new approach to performing the interventional electrophysiology procedure. The study population will consist of adult patients requiring ablation for type I atrial flutter.

Study subjects will require a follow-up visit or telephone call at 7 days post procedure.

Accordingly, the expected total study duration is approximately six months with study start planned for October 2014.

ELIGIBILITY:
Inclusion Criteria:

* First time indication for type I atrial flutter ablation
* Age 18 or above
* Patients willing and able (mentally and physically capable per physician's discretion) to understand the investigational nature, potential risks and benefits of the study and able to provide written informed consent to participate in the study and agree to comply with follow-up visits and evaluation
* Patients able to receive anticoagulation therapy to achieve adequate anticoagulation

Exclusion Criteria:

* Contraindication for MRI diagnostic exam
* A cardiac ablation or cardiac surgery within 90 days prior to enrollment
* Documented intracardiac thrombus, tumor, bleeding, clotting or other abnormality that precludes catheter introduction and placement
* Myocardial infarction within 60 days prior to enrollment
* Current unstable angina
* History of cerebrovascular event (within 180 days prior to enrollment)
* Patients with an ejection fraction less than or equal to 30% within 90 day prior to enrollment
* Permanent leads in or through the right atrium
* Clinically significant structural heart disease (including tricuspid valve regurgitation, tricuspid valve stenosis or other congenital heart disease) that would preclude catheter introduction and placement, as determined by the Investigator
* Uncompensated congestive heart failure (NYHA Class III or IV)
* Arrhythmia is secondary to electrolyte imbalance, thyroid disease, or other
* reversible or non-cardiovascular cause
* Known sensitivity to heparin or warfarin
* Active or systemic infection
* Any other significant uncontrolled or unstable medical condition (including but not limited to hypertension and diabetes)
* Women who are pregnant or plan to become pregnant within the course of their participation in the investigation or who are breastfeeding
* Life expectancy of less than 12 months
* Patients with prosthetic valves
* Contraindicated for transfemoral venous access
* Older than 75 years
* Current enrollment in any other clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events | 1 day
  To provide scientific evidence that the Vision Ablation Catheter is safe as measured by the incidence of device and procedure related serious adverse events (SAEs).

SECONDARY OUTCOMES:
Number of participants with successful ablation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Professor, Principal Investigator — Heart Center Leipzig
Locations (1):
- Heart Center Leipzig, Leipzig, Germany

REFERENCES:
- [Background] Sommer P, Grothoff M, Eitel C, Gaspar T, Piorkowski C, Gutberlet M, Hindricks G. Feasibility of real-time magnetic resonance imaging-guided electrophysiology studies in humans. Europace. 2013 Jan;15(1):101-8. doi: 10.1093/europace/eus230. Epub 2012 Jul 31. PMID 22849974
- [Background] Eitel C, Hindricks G, Grothoff M, Gutberlet M, Sommer P. Catheter ablation guided by real-time MRI. Curr Cardiol Rep. 2014 Aug;16(8):511. doi: 10.1007/s11886-014-0511-6. PMID 24952899
- [Background] Piorkowski C, Grothoff M, Gaspar T, Eitel C, Sommer P, Huo Y, John S, Gutberlet M, Hindricks G. Cavotricuspid isthmus ablation guided by real-time magnetic resonance imaging. Circ Arrhythm Electrophysiol. 2013 Feb;6(1):e7-10. doi: 10.1161/CIRCEP.112.973719. No abstract available. PMID 23424226
- [Result] Hilbert S, Sommer P, Gutberlet M, Gaspar T, Foldyna B, Piorkowski C, Weiss S, Lloyd T, Schnackenburg B, Krueger S, Fleiter C, Paetsch I, Jahnke C, Hindricks G, Grothoff M. Real-time magnetic resonance-guided ablation of typical right atrial flutter using a combination of active catheter tracking and passive catheter visualization in man: initial results from a consecutive patient series. Europace. 2016 Apr;18(4):572-7. doi: 10.1093/europace/euv249. Epub 2015 Aug 27. PMID 26316146